CLINICAL TRIAL: NCT03033576
Title: A Phase II Randomized Study of Nivolumab (NSC-748726) With Ipilimumab (NSC-732442) or Ipilimumab Alone in Advanced Melanoma Patients Refractory to an Anti-PD1 or Anti-PD-L1 Agent
Brief Title: Testing Treatment With Ipilimumab and Nivolumab Compared to Treatment With Ipilimumab Alone in Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00105; NCI-2017-00105 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1616 (Other: SWOG); S1616 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2017-01-26; First posted 2017-01-27 (Estimated); Results first posted 2023-05-01 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Melanoma of Unknown Primary; Mucosal Melanoma; Unresectable Cutaneous Melanoma; Unresectable Melanoma
MeSH Terms: interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ipilimumab) (Active Comparator): Patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab
- Arm II (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 30 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm II (nivolumab, ipilimumab)

SUMMARY:
This phase II trial studies how well ipilimumab with or without nivolumab work in treating patients with melanoma that is stage IV or stage III and cannot be removed by surgery. Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression free survival (PFS) of patients with advanced melanoma refractory to an anti-PD-1 or anti-PD-L1 agent, treated with combination therapy ipilimumab plus nivolumab versus ipilimumab alone.

SECONDARY OBJECTIVES:

I. To estimate difference in T-cell infiltrate between on-study biopsy samples of patients who respond to combination therapy (including confirmed and unconfirmed, complete and partial response per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1, in each treatment arm).

II. To evaluate the objective response rate (ORR), defined as confirmed complete or partial response per RECIST 1.1, in each treatment arm.

III. To evaluate the overall survival (OS) of patients in each treatment arm. IV. To evaluate the toxicity profile of patients in each treatment arm.

TRANSLATIONAL OBJECTIVES:

I. To assess the marginal prognostic value of baseline T-cell density, T-cell receptor (TCR) clonality, mutational load, messenger ribonucleic acid (mRNA) and other phenotypical expression levels, and circulating tumor deoxyribonucleic acid (DNA) in terms of response.

II. To assess the joint prognostic value of T-cell density, TCR clonality, and mutational load, mRNA and other phenotypical expression levels, and circulating tumor DNA in terms of response.

III. To identify T-cell poor subtype(s) that are associated with response.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ipilimumab intravenously (IV) over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 30 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years and then annually for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed melanoma that is either stage IV or unresectable stage III; patients may have primaries of cutaneous, mucosal or unknown origin; patients with uveal (ocular) primary are not eligible
* Patients must have measurable disease per RECIST 1.1; all measurable lesions must be assessed by physical examination, computed tomography (CT) scans or magnetic resonance imaging (MRI) within 28 days prior to registration; if the only measurable disease is cutaneous or subcutaneous, lesions must be at least 10 mm in greatest dimension and able to be serially recorded using calipers and photographs; tests used to assess non-measurable disease must have been performed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form
* Patients with central nervous system (CNS) metastases must have all lesions adequately treated with stereotactic radiation therapy, craniotomy, Gamma Knife (registered trademark) therapy, or whole brain radiotherapy, with no subsequent evidence of CNS progression; patients must not have required steroids for at least 14 days prior to registration; patients with a history of central nervous system metastases must have MRI of the brain within 42 days prior to registration
* Patients must have had prior treatment with anti-PD1 or anti-PD-L1 agents and had documented disease progression per the treating physician either while on these agents or after stopping therapy with these agents without intervening therapy; patients who received adjuvant therapy for previously resected disease with PD-1 or PD-L1 agents may also be eligible if disease recurrence occurred while still receiving the PD-1 or PD-L1 therapy and no intervening therapy was received; patients must have discontinued anti-PD-1 or anti-PD-L1 therapy at least 21 days prior to registration
* Patients must be >= 18 years of age
* Patients must have Zubrod performance status of =< 2
* Patients must have complete history and physical examination within 28 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500/mcL (within 28 days prior to registration)
* Hemoglobin >= 8 g/dL (within 28 days prior to registration)
* Platelets >= 100,000/mcL (within 28 days prior to registration)
* Total bilirubin =< 2.5 x institutional upper limit of normal (IULN) (except patients with Gilbert's syndrome) (within 28 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both =< 5 x IULN (within 28 days prior to registration)
* Serum creatinine =< 2.0 x IULN within 28 days prior to registration
* Patients with a known history of human immunodeficiency virus (HIV) must have CD4 count >= institutional lower limit of normal within 28 days prior to registration
* Patients with a known history of congestive heart failure (CHF), cardiomyopathy, myocarditis, myocardial infarction (MI), exposure to cardiotoxic medications, or with a clinical history suggestive of the above must have an electrocardiography (EKG) and echocardiogram (ECHO) performed within 42 days prior to registration and as clinically indicated while on treatment
* Patients with new symptoms of congestive heart failure (CHF), cardiomyopathy, myocarditis, myocardial infarction (MI), or exposure to cardiotoxic medications must have a cardiology consultation, creatinine phosphokinase (CPK), and troponin testing at prestudy and as clinically indicated
* Males who are sexually active with women of reproductive potential must have agreed to use birth control throughout the study and for 7 months after completion of protocol treatment; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (vasectomy); if at any point a previously celibate patient chooses to become heterosexually active during or within 7 months after completion of protocol treatment, he is responsible for beginning effective contraceptive measures
* Patients must submit archival tissue (if available) for translational medicine; patients must also be willing to undergo biopsies and submit tissue and blood for translational medicine
* Patients must be offered the opportunity to participate in specimen banking of leftover tissue for future research
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Exclusion Criteria:

* Patients must not have achieved a partial or complete response to the anti-PD-1 or anti-PD-L1 agents prior to progression per the treating physician
* Patients must not have had any systemic therapy, including anti-PD-1 or anti-PD-L1 agents, within 21 days prior to registration
* Patients must not have had prior radiation therapy within 14 days prior to registration
* Patients must not have had:

  * Prior treatment with ipilimumab or other CTLA-4 antagonists
  * Systemic therapy between progression on the anti-PD-1 or anti-PD-L1 agents and registration
  * Note: Systemic therapy (including BRAF-targeting agents) prior to anti-PD-1 or anti-PD-L1 therapy is allowed
* Patients must not be planning to require any additional form of systemic anti-tumor therapy while on protocol treatment
* Patients must not have known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection prior to registration
* Patients must not have an active infection requiring systemic therapy at time of registration
* Patients must not have organ allografts
* Patients must not have received systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days prior to registration; inhaled or topical steroids, and adrenal replacement doses =< 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease
* Patients must not have a history of immune-mediated pneumonitis or colitis that required interruption of therapy or treatment of steroids
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage 0, I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for two years
* Patients must not be pregnant or nursing due to risk of fetal or nursing infant harm; females of reproductive potential must have negative serum pregnancy test within 2 days prior to registration and agree to use an effective contraceptive method throughout the study and for 5 months after completion of protocol treatment; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; if at any point a previously celibate patient chooses to become heterosexually active during or within 5 months after protocol treatment, she is responsible for beginning effective contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2024-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari M Vanderwalde, Principal Investigator — SWOG Cancer Research Network
Locations (638):
- United States (638):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Stephens Memorial Hospital, Norway, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Hospital, Kalamazoo, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - The West Clinic - Corinth, Corinth, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Nebraska Medicine Heartland Hematology Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - The West Clinic - Wolf River, Germantown, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - The West Clinic - Mid-Town, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] VanderWalde A, Bellasea SL, Kendra KL, Khushalani NI, Campbell KM, Scumpia PO, Kuklinski LF, Collichio F, Sosman JA, Ikeguchi A, Victor AI, Truong TG, Chmielowski B, Portnoy DC, Chen Y, Margolin K, Bane C, Dasanu CA, Johnson DB, Eroglu Z, Chandra S, Medina E, Gonzalez CR, Baselga-Carretero I, Vega-Crespo A, Garcilazo IP, Sharon E, Hu-Lieskovan S, Patel SP, Grossmann KF, Moon J, Wu MC, Ribas A. Ipilimumab with or without nivolumab in PD-1 or PD-L1 blockade refractory metastatic melanoma: a randomized phase 2 trial. Nat Med. 2023 Sep;29(9):2278-2285. doi: 10.1038/s41591-023-02498-y. Epub 2023 Aug 17. PMID 37592104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 94 participants were assessed for eligibility; 24 to the Ipilimumab arm and 70 to the Nivolumab + Ipilimumab arm. Two participants were deemed ineligible, leaving 92 eligible and analyzable participants.
Groups:
- Ipilimumab: Active Comparator: Arm I (ipilimumab)
  Patients receive ipilimumab 3mg/kg IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
- Nivolumab + Ipilimumab: Experimental: Arm II (nivolumab, ipilimumab)
  Patients receive nivolumab 1 mg/kg IV over 30 minutes and ipilimumab 3 mg/kg IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab 480 mg IV over 30 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Ipilimumab | Nivolumab + Ipilimumab
Started | 24 | 70
Eligible | 23 | 69
Received Protocol-directed Therapy | 23 | 68
Completed | 8 | 0
Not Completed | 16 | 70
Not completed — Ineligible | 1 | 1
Not completed — Adverse Event | 4 | 20
Not completed — Progression/relapse | 9 | 36
Not completed — Death | 1 | 1
Not completed — Patient refusal | 1 | 6
Not completed — Other, unspecified reasons | 0 | 4
Not completed — Currently on protocol therapy | 0 | 2

BASELINE CHARACTERISTICS:
Population: Only eligible participants were assessed for baseline measures.
Groups:
- Ipilimumab: Active Comparator: Arm I (ipilimumab)
  Patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
- Nivolumab + Ipilimumab: Experimental: Arm II (nivolumab, ipilimumab)
  Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 30 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Ipilimumab | Nivolumab + Ipilimumab | Total
Number analyzed (Participants) | 23 | 69 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 35 | 44
  >=65 years | 14 | 34 | 48
Age, Continuous [Median (Full Range); unit: years] | 69 [40 to 91] | 64 [34 to 90] | 67 [34 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 23 | 31
  Male | 15 | 46 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 63 | 85
  Black | 0 | 1 | 1
  Asian | 1 | 3 | 4
  Unknown | 0 | 2 | 2
Zubrod Performance Status Score [Count of Participants; unit: Participants] — Zubrod performance status scores range from 0 to 2, with higher scores reflecting greater disability.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    0 | 15 | 45 | 60
    1 | 6 | 20 | 26
    2 | 2 | 4 | 6
LDH [Count of Participants; unit: Participants] — Blood lactate dehydrogenase (LDH) levels were measured and classified as either elevated or normal.
  Participants
    Elevated | 6 | 9 | 15
    Normal | 5 | 28 | 33
    LDH Not Done | 12 | 32 | 44
AJCC Melanoma Classification [Count of Participants; unit: Participants] — Participants' disease stage was classified according to the AJCC melanoma classification. Stage III: Any T, N3, M0. Stage IV: Any T, Any N, M1.
  Participants
    Stage III | 6 | 12 | 18
    Stage IV | 17 | 57 | 74
Prior Adjuvant Therapy [Count of Participants; unit: Participants]
  No prior adjuvant therapy | 17 | 58 | 75
  Adjuvant PD-1 | 3 | 7 | 10
  Adjuvant BRAF/MEK | 0 | 2 | 2
  Other Adjuvant Therapy | 3 | 2 | 5
Prior Metastatic Therapy [Count of Participants; unit: Participants]
  Adjuvant Therapy Only | 1 | 6 | 7
  Anti-PD-1 only | 20 | 54 | 74
  BRAF/MEK followed by PD-1 | 1 | 1 | 2
  Other anti-PD-1 combination | 1 | 8 | 9
Duration of prior anti-PD1/PD-L1 Therapy [Count of Participants; unit: Participants]
  < 6 Months | 15 | 44 | 59
  >= 6 Months | 8 | 25 | 33

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the time from date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Participants last known to be alive without report of progression are censored at date of last contact. Progression is defined as either 20% increase in the sum of diameters of target measurable lesions, unequivocal progression of non-measurable disease in the opinion of the treating physician, appearance of any new lesion, or death due to disease without prior documentation of progression and without symptomatic deterioration. Symptomatic deterioration is defined as global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years
Population: Only eligible participants were analyzed for PFS.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Ipilimumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 23 | 69
months | 2.7 [2.5 to 2.9] | 3.1 [2.8 to 5.3]
Statistical Analysis 1: Comparison: Ipilimumab vs Nivolumab + Ipilimumab; The statistical design assumed exponential PFS with a median of 3.0 months on the ipilimumab group (null hypothesis). The study was powered to detect a change in median PFS to 6.0 months in the combination therapy group (corresponding to an HR of 0.50). A total of 84 participants (63 randomized to combination group and 21 to ipilimumab group) with 78 events (across both groups) would provide 89% power for a one-sided alpha of 10% using a log-rank test; Test type: Superiority; p = 0.04, Log Rank — Pre-specified one-sided alpha=0.1; Hazard Ratio (HR) = 0.63, 90% CI 2-sided [0.41 to 0.97]

2. Secondary Outcome: Change in CD8+ Expression
Description: Will estimate the quantitative change in CD8+ expression from baseline to day 28 on-study between patients who eventually respond and patients who do not respond in the Nivolumab + Ipilimumab arm.
Time Frame: Up to 3 years
Population: There were 83 total participants with biopsies available; 76 with a baseline biopsy and 56 with a biopsy from 28 days after start of protocol therapy. This resulted in a total of 40 paired biopsies on both arms after excluding samples that could not be analyzed because of absence of tumor due or insufficient tumor cells. Our analysis population for this outcome measure includes the 29 participants on the combination Nivolumab + Ipilimumab arm that had an analyzable paired biopsy.
Measure: Mean (Standard Deviation); unit: log10[cells per mm^2]
Groups:
- Responders; Non-Responders: Participants on the combination Nivolumab + Ipilimumab arm that responded to protocol therapy.
- Overall: All participants on the combination Nivolumab + Ipilimumab arm that were had biopsies available at baseline and four weeks after the start of protocol therapy.
Arm/Group | Responders | Non-Responders | Overall
Number analyzed (Participants) | 12 | 17 | 29
log10[cells per mm^2] | 0.4291 (0.821187) | 0.2585 (0.550321) | 0.3291 (0.667305)

3. Secondary Outcome: Overall Objective Response Rate
Description: The overall objective response rate is defined as percentage of participants that achieved confirmed and unconfirmed, complete and partial responses. Complete response is defined as complete disappearance of all target and non-target lesions, no new lesions, and no disease related symptoms. Partial response applies only to patients with at least one measurable lesion and is defined as >= 30% decrease of the sum of diameters of all target measurable lesions, no unequivocal progression of non-measurable disease, and no new lesions.
Time Frame: Up to 3 years
Population: All eligible participants were considered analyzable for this endpoint.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 23 | 69
percentage of participants | 9 [2 to 25] | 28 [19 to 38]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to the date of death from any cause.
Time Frame: Up to 3 years
Population: All eligible participants were included in the overall survival analysis.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Ipilimumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 23 | 69
months | 14.5 [8.1 to NA] — There was insufficient follow-up data to estimate an upper limit. | 22.1 [15.4 to 32.4]
Statistical Analysis 1: Comparison: Ipilimumab vs Nivolumab + Ipilimumab; Test type: Superiority; p = 0.28, Log Rank; Hazard Ratio (HR) = 0.83, 90% CI 2-sided [0.50 to 1.39]

5. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported. Adverse Events (AEs) are reported by CTCAE Version 4.0.
Time Frame: Duration of treatment and follow-up until death or 3 years post registration
Population: Participants who received at least one dose of protocol treatment
Measure: Number; unit: Participants
Arm/Group | Ipilimumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 23 | 68
Participants
  Acute kidney injury | 0 | 1
  Adrenal insufficiency | 1 | 3
  Alanine aminotransferase increased | 2 | 5
  Alkaline phosphatase increased | 1 | 2
  Anemia | 0 | 4
  Anorexia | 0 | 2
  Arthralgia | 0 | 1
  Aspartate aminotransferase increased | 2 | 5
  Atrial fibrillation | 1 | 1
  Autoimmune disorder | 0 | 1
  Blood bilirubin increased | 1 | 0
  Colitis | 0 | 3
  Colonic perforation | 1 | 0
  Dehydration | 1 | 1
  Diarrhea | 3 | 9
  Disseminated intravascular coagulation | 0 | 1
  Endocrine disorders - Other, specify | 0 | 3
  Enterocolitis | 0 | 1
  Fatigue | 2 | 4
  Fever | 0 | 1
  Hyperglycemia | 1 | 0
  Hypernatremia | 0 | 1
  Hypocalcemia | 0 | 1
  Hypokalemia | 0 | 3
  Hyponatremia | 1 | 4
  Hypophosphatemia | 1 | 0
  Hypotension | 0 | 4
  Hypothyroidism | 0 | 1
  Infections and infestations - Other, specify | 0 | 1
  Lung infection | 0 | 1
  Lymphocyte count decreased | 0 | 2
  Metabolism and nutrition disorders - Other, specify | 0 | 1
  Nausea | 0 | 2
  Pain | 0 | 2
  Pruritus | 0 | 3
  Rash maculo-papular | 1 | 4
  Syncope | 0 | 1
  Uveitis | 0 | 1
  Vomiting | 0 | 3

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow-up until death or 3 years post registration
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only eligible participants who received protocol treatment were evaluated for adverse events (91 total; 23 on the ipilimumab arm; 68 on the nivolumab + ipilimumab arm), whereas all eligible participants were evaluated for all-cause mortality (92 total; 23 on the ipilimumab arm; 69 on the nivolumab + ipilimumab arm).
Arm/Group | Ipilimumab | Nivolumab + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 14/23 | 40/69
Serious Adverse Events (participants affected / at risk) | 10/23 | 38/68
Other Adverse Events (participants affected / at risk) | 23/23 | 66/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=23) | Nivolumab + Ipilimumab (N=68)
Anemia (Blood and lymphatic system disorders) | 0 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Heart failure (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 3
Endocrine disorders-Other (Endocrine disorders) | 0 | 3
Hypothyroidism (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Bloating (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 4
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 8
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 4
Chills (General disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 0 | 3
Flu like symptoms (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Autoimmune disorder (Immune system disorders) | 0 | 1
Esophageal infection (Infections and infestations) | 0 | 1
Infections and infestations-Other (Infections and infestations) | 1 | 3
Lung infection (Infections and infestations) | 0 | 4
Sepsis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 3
Alkaline phosphatase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 4
Blood bilirubin increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1
GGT increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 4
Thromboembolic event (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=23) | Nivolumab + Ipilimumab (N=68)
Anemia (Blood and lymphatic system disorders) | 6 | 22
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 | 4
Sinus tachycardia (Cardiac disorders) | 1 | 7
Adrenal insufficiency (Endocrine disorders) | 1 | 6
Endocrine disorders-Other (Endocrine disorders) | 0 | 4
Hyperthyroidism (Endocrine disorders) | 0 | 4
Hypothyroidism (Endocrine disorders) | 2 | 6
Blurred vision (Eye disorders) | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 9
Constipation (Gastrointestinal disorders) | 4 | 13
Diarrhea (Gastrointestinal disorders) | 9 | 24
Dry mouth (Gastrointestinal disorders) | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 5
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 6
Mucositis oral (Gastrointestinal disorders) | 1 | 5
Nausea (Gastrointestinal disorders) | 11 | 23
Vomiting (Gastrointestinal disorders) | 5 | 10
Chills (General disorders) | 2 | 6
Edema limbs (General disorders) | 3 | 8
Fatigue (General disorders) | 13 | 35
Fever (General disorders) | 3 | 12
Flu like symptoms (General disorders) | 0 | 4
Non-cardiac chest pain (General disorders) | 2 | 4
Pain (General disorders) | 2 | 10
Autoimmune disorder (Immune system disorders) | 2 | 0
Infections and infestations-Other (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 2 | 5
Alanine aminotransferase increased (Investigations) | 4 | 20
Alkaline phosphatase increased (Investigations) | 6 | 11
Aspartate aminotransferase increased (Investigations) | 5 | 22
Blood bilirubin increased (Investigations) | 0 | 8
Creatinine increased (Investigations) | 4 | 9
Investigations-Other (Investigations) | 1 | 8
Lymphocyte count decreased (Investigations) | 4 | 11
Platelet count decreased (Investigations) | 2 | 1
Weight loss (Investigations) | 3 | 9
White blood cell decreased (Investigations) | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 4 | 22
Dehydration (Metabolism and nutrition disorders) | 3 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 9
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 16
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 8
Hyponatremia (Metabolism and nutrition disorders) | 7 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 9
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 5
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 14
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Dizziness (Nervous system disorders) | 0 | 12
Dysgeusia (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 6 | 19
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 6
Anxiety (Psychiatric disorders) | 2 | 3
Depression (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 2 | 6
Renal and urinary disorders-Other (Renal and urinary disorders) | 0 | 6
Urinary frequency (Renal and urinary disorders) | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 28
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 25
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 12
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 4
Hot flashes (Vascular disorders) | 1 | 4
Hypertension (Vascular disorders) | 2 | 12
Hypotension (Vascular disorders) | 2 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03033576/Prot_SAP_000.pdf